CLINICAL TRIAL: NCT00092430
Title: A Comparison of the Safety, Tolerability, and Immunogenicity of a Refrigerator-Stable Measles, Mumps, Rubella, and Varicella Combination Vaccine V221 (Refrigerated) Versus V221 (Frozen) in Healthy Children
Brief Title: Study to Evaluate Frozen Versus Refrigerated MMRV (Combined Measles, Mumps, Rubella, and Varicella) Investigational Vaccine (V221-016)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V221-016; 2004_076
Record Dates: First submitted 2004-09-22; First posted 2004-09-27 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Measles; Mumps; Rubella; Varicella
MeSH Terms: conditions — Measles; Mumps; Rubella; Chickenpox | interventions — Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Biological: V221, measles, mumps, rubella and varicella (Oka/Merck) virus vaccine live / Duration of Treatment: 12 weeks

SUMMARY:
The purpose of this study is to demonstrate that an investigational refrigerated vaccine with measles, mumps, rubella, and varicella is well tolerated and has similar immune response when compared to a frozen vaccine with measles, mumps, rubella, and varicella.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children 12-23 months of age

Exclusion Criteria:

* Previously had measles, mumps, rubella, or varicella
* Compromised immune system

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200
Dates: Start 2002-09-26 (Actual); Primary Completion 2003-06-09 (Actual); Study Completion 2003-06-09 (Actual)

PRIMARY OUTCOMES:
Percent of patients demonstrating adequate antibody titers 6 weeks following administration

SECONDARY OUTCOMES:
Geometric mean titers (GMT) 6 weeks post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Bernstein HH, Eves K, Campbell K, Black SB, Twiggs JD, Reisinger KS, Conti RM, Flodmark CE, Rombo L, Klopfer S, Schodel F, Hartzel J, Kuter BJ; Refrigerator-Stable Formulation Study Group for ProQuad. Comparison of the safety and immunogenicity of a refrigerator-stable versus a frozen formulation of ProQuad (measles, mumps, rubella, and varicella virus vaccine live). Pediatrics. 2007 Jun;119(6):e1299-305. doi: 10.1542/peds.2006-2283. Epub 2007 May 14. PMID 17502347
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html